CLINICAL TRIAL: NCT02683356
Title: Optical Coherence Tomography to Improve Outcome for Coronary Revascularisation Using Bioresorbable Vascular Scaffolds
Acronym: OPTICO-BVS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company stopped selling BVS/ No 5 year FUP will be done
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016-01-16
Record Dates: First submitted 2016-01-22; First posted 2016-02-17 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Coronary Occlusion
Keywords: Percutaneous Coronary Intervention; Stents
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCT-guided PCI (Active Comparator): OCT before and after Stent implantation
  Interventions: Other: OCT-guided PCI
- Angiography-guided PCI (Active Comparator): OCT after Stent implantation
  Interventions: Other: Angiography-guided PCI

INTERVENTIONS:
Other: OCT-guided PCI — Patients assigned to the OCT-guided PCI strategy will undergo OCT prior to PCI to determine vessel and lesion dimensions and treatment strategy. OCT will be repeated at the end of the procedure and corrective PCI will aim to optimize the PCI result according to pre-specified criteria in terms of minimal lumen area, scaffold expansion, apposition, residual dissections or intra-scaffold thrombus formation
  Arms: OCT-guided PCI
Other: Angiography-guided PCI — Patients assigned to the OCT-guided PCI strategy will only undergo OCT after PCI to determine vessel and lesion dimensions and treatment strategy.
  Arms: Angiography-guided PCI

SUMMARY:
Fully Bioresorbable Vascular Scaffolds (BVS) have been introduced with the objective to preserve native vessel geometry, allow for adaptive vessel remodeling with late lumen gain, restore physiological vasomotion, and avoid late adverse events including restenosis and scaffold thrombosis. Although randomized clinical trials in low risk patients to date suggest non-inferiority in terms of safety and efficacy compared with metallic DES, several reports have raised concerns regarding the scaffold thrombosis highlighting the importance of technical considerations regarding lesion preparation and scaffold expansion. OCT offers the opportunity to plan the procedure and optimize the implantation of BVS.

The hypothesis of the present study is that a strategy of OCT-guided PCI using BVS is superior to angiography-guided PCI (e.g. by selecting scaffold dimension on the basis of a pre-procedural OCT and applying corrective measures in case of suboptimal treatment result as indicated by OCT).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patient provides signed written informed consent before any study-specific procedure.
3. De novo native coronary artery disease with lesions that have a distal and proximal reference vessel diameter in the range between 2.25mm and 3.8mm.
4. Single or multi vessel disease. For multi vessel disease up to two vessels and three lesions treated at baseline with no more than two lesions per vessel. Vessel is defined as, left anterior descending, left circumflex, and right coronary arteries. Any branch within the vessel is considered part of the vessel.
5. Full revascularization of all lesions should be achievable (staged PCI not recommended)
6. Elective or ad hoc PCI, stable angina and acute coronary syndrome (NSTE-ACS and STEMI).
7. Angiographically significant (>50% visual estimation) stenosis present in at least one native coronary artery and evidence of ischemia.

Exclusion Criteria:

1. Subjects with left main lesion.
2. Aorto-ostial lesion location within 3 mm of the aorta junction (both right and left).
3. Subjects with restenosis or stent thrombosis in the target vessel.
4. Severely calcified lesions requiring rotablation.
5. Bifurcation with sidebranch >2.5mm or any sidebranch that possibly requires treatment with angulation >70°
6. Severe angulation (>90°) or excessive tortuosity (>two 45° angles)
7. Known renal insufficiency (serum creatinine clearance <45ml/min or receiving dialysis).
8. Vessel(s) and lesion(s) not amenable for PCI, for example diffuse disease.
9. Female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy
10. Life expectancy less than 1 year.
11. Indication for oral anticoagulation
12. Known allergy against protocol-required medications including ASA, prasugrel, ticagrelor, clopidogrel, heparin, iodinated contrast (the latter in case it cannot be adequately premedicated)
13. History of bleeding diathesis or known coagulopathy.
14. Planned surgery within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Minimal in-scaffold lumen area (mm2) as assessed by OCT | 6 months
  The lumen area is assessed by OCT

SECONDARY OUTCOMES:
Number of adverse events | 6 months
  Adverse events are defined as scaffold underexpansions, significant strut malappositions or uncovered struts, expansion asymmetries, any intrascaffold tissue, edge dissections, or restenoses (as assessed by OCT)
OCT imaging endpoints | 6 months
  Scaffold underexpansion, significant strut malapposition or uncovered struts, expansion asymmetry, any intrascaffold tissue, edge dissection, or restenosis. (as assessed by OCT)
Additional OCT imaging endpoints | 6 months
  * Significant malapposed scaffold struts, %
  * Malapposed scaffold struts, %
  * Uncovered scaffold struts, %
  * Incomplete scaffold apposition area, mm2
  * Incomplete scaffold apposition distance, mm
  * Neointimal thickness, µm
  * Neointimal area, mm2
  * Volume obstruction, %
OCT imaging endpoints | end of procedure
  * Minimal in-scaffold lumen area, mm
  * Scaffold expansion, %
  * No of patients with scaffold expansion <80%
  * % lesions with significant malapposition
  * % malapposed struts
angiographic endpoints | end of procedure
  * acute lumen gain
  * in-scaffold minimal lumen diameter
  * in-segment minimal lumen diameter
  * in-scaffold % diameter stenosis
  * in-segment % diameter stenosis
angiographic endpoints | 6 months
  * In-scaffold late lumen loss, mm
  * In-segment late lumen loss, mm
  * In-scaffold % diameter stenosis
  * In-segment % diameter stenosis
  * Binary restenosis, %
  * Percent diameter stenosis, %

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, MD PhD, Study Chair — Bern University Hospital, Switzerland; Stephan Windecker, Prof. MD, Principal Investigator — Bern University Hospital, Switzerland
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No